CLINICAL TRIAL: NCT00582335
Title: Identification of New Colorectal Cancer Genes
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 98-003
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Genetic testing; Genetic mutations
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Tissue (tumor)

SUMMARY:
The purpose of this study is to define new genes for family risks of developing colon cancer.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most significant causes of cancer morbidity and mortality in the United States. In 1997, approximately 130,000 men and woman were diagnosed with colorectal cancer (fourth most common cancer site) and approximately 55,000 died of this disease (second most common cause of cancer deaths); (Cancer Facts & Figures, 1997).

Genetic factors clearly contribute to the etiology of colorectal cancer. Because there is evidence to suggest genetically determined susceptibility to colorectal cancer exists in a proportion of newly diagnosed cases each year, we are conducting a study to identify new genes that are associated with an increased susceptibility to familial colorectal cancer by analysis of families with a clustering of colorectal cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Able to provide informed consent
* Any family in which a minimum of two first-degree relatives either are, or have previously been, affected with primary colorectalcancer. These "minimum inclusion criteria" must be met within three generations of the proband or kindreds in which colorectal cancer and lymphoma or renal cell cancer are present or in kindreds in which lymphoma alone or lymphoma and renal cell cancer are present

Exclusion Criteria:

* Age less than 18 years
* Family not at increased risk for familial colorectal cancer (see Section 4.1)
* Family with a hereditary polyposis syndrome (e.g. classic FAP)
* Not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: families seen at MSKCC with at least two first-degree relatives affected with colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 1998-02-10 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Evidence of mutations in selected candidate genes | 10 years 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org